CLINICAL TRIAL: NCT03565679
Title: SpO2 Accuracy Comparison of Medline ReNewal Sensors to Arterial Blood CO-Oximetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medline Industries (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: PR 2018-268
Record Dates: First submitted 2018-05-09; First posted 2018-06-21 (Actual); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Arterial Oxygen Saturation; Healthy

STUDY DESIGN:
Intervention Model Description: Subjects will recline for the study. Reference sensors will be placed on each subject to evaluate the SpO2 accuracy and performance. Shield material may be used between any adjacent finger sensors to prevent optical crosstalk. Simultaneous data collection will be set up for devices under test. The data from the test devices will be collected by the sponsor or trained Clinimark Study staff. Data will be collected for 1 second intervals data analysis. The SpO2 accuracy of the test devices will be evaluated over the oxygen saturation range between 70-100%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Masimo SpO2 Adhesive Sensors, Adtx (1859) & (2329) (Experimental): Reference sensors from the reprocessed oximeter device will be placed on each subject to evaluate the SpO2 accuracy and performance.
  Interventions: Device: MEDLINE RENEWAL PULSE OXIMETRY SENSORS
- Covidien Nellcor SpO2 Sensor, MAX-A and MAX-N (Sham Comparator): A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.
  Interventions: Device: CO-OXIMETRY SENSORS

INTERVENTIONS:
Device: MEDLINE RENEWAL PULSE OXIMETRY SENSORS — An oximeter is a device used to transmit radiation at a known wavelength(s) through blood and to measure the blood oxygen saturation based on the amount of reflected or scattered radiation. Pulse oximetry monitoring is considered a standard physiological measurement and is used by clinicians in everyday situations to estimate arterial oxygen saturation. Because an arterial sample of blood is not required to make the measurement, the pulse oximeter can provide non-invasive real time information.
  Arms: Masimo SpO2 Adhesive Sensors, Adtx (1859) & (2329)
Device: CO-OXIMETRY SENSORS — A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.
  Arms: Covidien Nellcor SpO2 Sensor, MAX-A and MAX-N

SUMMARY:
The purpose of this clinical study is to validate the SpO2 accuracy of the Medline ReNewal pulse oximetry sensors during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. The end goal is to provide supporting documentation for the SpO2 accuracy validation of the ReNewal sensors.

It is required that the Accuracy Root Mean Square (ARMS) performance of the ReNewal pulse oximetry sensors will meet a specification of 3 or better in non-motion conditions for the range of 70 - 100% SaO2 thereby demonstrating an acceptable SpO2 accuracy performance specification.

DETAILED DESCRIPTION:
An oximeter is a device used to transmit radiation at a known wavelength(s) through blood and to measure the blood oxygen saturation based on the amount of reflected or scattered radiation. Pulse oximetry monitoring is considered a standard physiological measurement and is used by clinicians in everyday situations to estimate arterial oxygen saturation. Because an arterial sample of blood is not required to make the measurement, the pulse oximeter can provide non-invasive real time information. The clinical use of pulse oximeters has reduced the frequency and necessity of invasive arterial blood sampling and has helped to improve patient safety by providing continuous information to clinicians about patients' oxygenation status.

The Medline ReNewal Reprocessed pulse oximeter sensors are indicated for single patient use when continuous noninvasive arterial oxygen saturation and pulse rate monitoring are required. Following clinical use, each sensor is returned to Medline ReNewal where it is cleaned, disinfected, and packaged for an additional clinical use. Each sensor is tracked through the reprocessing cycle to monitor the number of times the sensor has been reprocessed. The purpose of this study will be to test the accuracy of the SpO2 component of the devices.

The SpO2 accuracy performance of ReNewal pulse oximetry sensors will be evaluated during non-motion conditions over the range of 70-100% SaO2 and compared to arterial blood samples assessed by CO-Oximetry. A minimum of 10 healthy adult subjects, ranging in pigmentation from light to dark, will be enrolled in the study to meet the study design requirements defined by International Organization for Standardization (ISO) 80601-2-61:2011 and by the FDA's Guidance for Pulse Oximeters (March 4, 2013). The subjects will have an arterial catheter placed in the radial artery to allow for simultaneous blood samples during stable plateaus of induced hypoxic levels. The investigational devices will be placed on the fingers of both hands for the test sites per the instructions for use. Simultaneous data collection will be set up for each of the systems under test. For the data analysis, the control oximeter will be used to assess the stability of each data point. Data that is found to be unstable will be removed prior to the comparative analysis. Next the CO-Oximeter data will be reviewed to make sure it does not contain any anomalous values such as elevated, low or inconsistent carboxyhemoglobin (COHb), methemoglobin (MetHb), or total hemoglobin (tHb) data. Anomalous values will be removed from the analysis prior to pairing of the SpO2 and SaO2 data. The Accuracy Root Mean Square (ARMS) calculation is used to determine the SpO2 accuracy performance. Success will be achieved with an ARMS of 3 or better showing equivalence to the Gold Standard Reference CO-Oximetry providing documentation to support SpO2 accuracy claims for the investigational device(s).

The study population will include 10-15 healthy non-smoking (or has refrained from smoking for 2 days) competent adults 18-50 years of age. The subject selection will be an equitable distribution of males and females of any race with varying skin tones including at least 2 darkly pigmented subjects or 15% of the subject pool, whichever is larger. Data collection will occur over a 2-5 day period for this study population. Follow-up with each subject will be conducted within 5 days following participation in the study and will be conducted via telephone, text or email.

ELIGIBILITY:
Inclusion Criteria:

* 10-15 Adults with a minimum of 3 males and a minimum of 3 females, with the balance made up of either
* Subject must have the ability to understand and provide written informed consent
* Subject is 18 to 50 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker or who has not smoked within 2 days prior to the study

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Females who are pregnant, who are trying to get pregnant, or have a urine test positive for pregnancy on the day of the study
* Smoker Subjects who have refrained will be screened for COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Subjects with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, chronic obstructive pulmonary disease (COPD), lung disease
* Subjects with known heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * hypertension: systolic >140mmHg, Diastolic >90mmHg on 3 consecutive readings (reviewed during health screen).
  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form (self-reported)

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury
  * cancer / chemotherapy
* Subjects with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Subjects with prior or known allergies to iodine or lidocaine (or similar pharmacological agents, e.g. Novocaine)
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test
* Unwillingness or inability to remove colored nail polish from test digits.
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Avista Adventist Hospital, Staff Anesthesiologist
Locations (1):
- Clinimark Desaturation Laboratory, Site ID# 001, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- MEDLINE RENEWAL PULSE OXIMETRY and Reference CO-oximetery: Reference sensors from the reprocessed oximeter device will be placed on each subject to evaluate the SpO2 accuracy and performance.
  Reprocessed Oximeter: is a device used to transmit radiation at a known wavelength(s) through blood and to measure the blood oxygen saturation based on the amount of reflected or scattered radiation. Pulse oximetry monitoring is considered a standard physiological measurement and is used by clinicians to estimate arterial oxygen saturation. Because an arterial sample of blood is not required to make the measurement, the pulse oximeter can provide non-invasive real time information.
  Whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.
  Reference Oximeter: A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.
Period: Overall Study
Arm/Group | MEDLINE RENEWAL PULSE OXIMETRY and Reference CO-oximetery
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MEDLINE RENEWAL PULSE OXIMETRY& Reference CO-oximetry Sensors: Reference sensors from the reprocessed oximeter device will be placed on each subject to evaluate the SpO2 accuracy and performance.
  Reprocessed Oximeter: is a device used to transmit radiation at a known wavelength(s) through blood and to measure the blood oxygen saturation based on the amount of reflected or scattered radiation. Pulse oximetry monitoring is considered a standard physiological measurement and is used by clinicians to estimate arterial oxygen saturation. Because an arterial sample of blood is not required to make the measurement, the pulse oximeter can provide non-invasive real time information.
  A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.
  Reference Oximeter: A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.
Arm/Group | MEDLINE RENEWAL PULSE OXIMETRY& Reference CO-oximetry Sensors
Number analyzed (Participants) | 10
Age, Continuous [Median (Standard Deviation); unit: years] | 27.58 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: SpO2 Percentage Specification
Description: Percentage of SpO2 (oxygen saturation by pulse oximetry) measured by the Reprocessed Oximeter pulse oximetry sensors during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry.
  The Accuracy root mean square (ARMS) between measured SpO2 and reference SaO2 (arterial oxygen saturation) must meett the 3% specification for each Medline Renewal Reprocessed pulse oximetry sensor style.
Time Frame: 2 hours
Population: Over 70 - 100% an ARMS ≤ 3% in non-motion conditions - Pass result
Measure: Number; unit: Percentage of SpO2
Groups:
- Masimo SpO2 Adhesive Sensors, Adtx (1859): Medline ReNewal Reprocessed Masimo SpO2 Adhesive Sensors, Adtx (1859) compared to Reference CO-Oximetry (functional SaO2)
- Masimo SpO2 Adhesive Sensors, Neo (2329): Medline ReNewal Reprocessed Masimo SpO2 Adhesive Sensors, Neo (2329)Comparison to Reference CO-Oximetry (functional SaO2)
- Covidien Nellcor SpO2 Sensor, MAX-A: Medline ReNewal Reprocessed Covidien Nellcor SpO2 Sensor, MAX-AComparison to Reference CO-Oximetry (functional SaO2)
- Covidien Nellcor SpO2 Sensor, MAX-N: Medline ReNewal Reprocessed Covidien Nellcor SpO2 Sensor, MAX-N Comparison to Reference CO-Oximetry (functional SaO2)
Arm/Group | Masimo SpO2 Adhesive Sensors, Adtx (1859) | Masimo SpO2 Adhesive Sensors, Neo (2329) | Covidien Nellcor SpO2 Sensor, MAX-A | Covidien Nellcor SpO2 Sensor, MAX-N
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percentage of SpO2 | 1.8 | 1.7 | 1.6 | 1.7

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- All Participants: All participants used every device
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03565679/Prot_SAP_000.pdf